CLINICAL TRIAL: NCT00653614
Title: A Multi-center, Double-blind, Randomized, Parallel-group Study to Evaluate Cycle Control and Safety of 6 Different Regimens of an Oral Contraceptive Containing Estradiol and Drospirenone in Healthy Female Volunteers Aged Between 18 and 35 Years Over 7 Cycles
Brief Title: Cycle Control and Safety of E2-DRSP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91765; 2007-005258-22 (EudraCT Number); 311926 (Other: Company Internal)
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Contraceptive, Oral, Hormonal
Keywords: Oral contraception
MeSH Terms: interventions — drospirenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): E2/DRSP (BAY 86-4891) dose 1 (SHT04984E) for 24 days and DRSP (ZK 30595) dose 1 (SHT04984F) for one day and placebo for three days in a 28 day cycle
  Interventions: Drug: E2/DRSP (BAY 86-4891) dose 1 (SH T04984E); Drug: DRSP (ZK 30595) dose 1 (SH T04984F); Drug: Placebo
- Arm 2 (Experimental): E2/DRSP (BAY 86-4891) dose 1 (SHT04984E) for 24 days and DRSP (ZK 30595) dose 1 (SHT04984F) for two days and placebo for two days in a 28 day cycle
  Interventions: Drug: E2/DRSP (BAY 86-4891) dose 1 (SH T04984E); Drug: DRSP (ZK 30595) dose 1 (SH T04984F); Drug: Placebo
- Arm 3 (Experimental): E2/DRSP (BAY 86-4891) dose 2 (80458739) for days 1-8, E2/DRSP (BAY 86-4891) dose 1 (SHT04984E) for days 9-16, E2/DRSP (BAY 86-4891) dose 3 (80458755) for days 17-24, and placebo for days 25-28 in a 28 day cycle
  Interventions: Drug: E2/DRSP (BAY 86-4891) dose 1 (SH T04984E); Drug: E2/DRSP (BAY 86-4891) dose 2 (80458739); Drug: E2/DRSP (BAY 86-4891) dose 3 (80458755); Drug: Placebo
- Arm 4 (Experimental): E2/DRSP (BAY 86-4891) dose 2 (80458739) for days 1-8, E2/DRSP (BAY 86-4891) dose 1 (SHT04984E) for days 9-16, E2/DRSP (BAY 86-4891) dose 3 (80458755) for days 17-24, placebo for 3 days, and DRSP (ZK 30595) dose 1 (SHT04984F) for one day in a 28 day cycle
  Interventions: Drug: E2/DRSP (BAY 86-4891) dose 1 (SH T04984E); Drug: E2/DRSP (BAY 86-4891) dose 2 (80458739); Drug: E2/DRSP (BAY 86-4891) dose 3 (80458755); Drug: E2/DRSP (BAY 86-4891) dose 4 (80458720); Drug: DRSP (ZK 30595) dose 1 (SH T04984F); Drug: Placebo
- Arm 5 (Experimental): E2/DRSP (BAY 86-4891) dose 2 (80458739) for days 1-8, E2/DRSP (BAY 86-4891) dose 4 (80458720) for days 9-16, E2/DRSP (BAY 86-4891) dose 5 (80458712) for days 17-24, and placebo for 4 days in a 28 day cycle
  Interventions: Drug: E2/DRSP (BAY 86-4891) dose 2 (80458739); Drug: E2/DRSP (BAY 86-4891) dose 5 (80458712); Drug: Placebo
- Arm 6 (Experimental): E2/DRSP (BAY 86-4891) dose 2 (80458739) for days 1-8, E2/DRSP (BAY 86-4891) dose 4 (80458720) for days 9-16, E2/DRSP (BAY 86-4891)dose 5 (80458712) for days 17-24, placebo for 3 days, and DRSP (ZK 30595) dose 2 (80458690) for one day in a 28 day cycle
  Interventions: Drug: E2/DRSP (BAY 86-4891) dose 2 (80458739); Drug: E2/DRSP (BAY 86-4891) dose 4 (80458720); Drug: E2/DRSP (BAY 86-4891) dose 5 (80458712); Drug: DRSP (ZK 30595) dose 2 (80458690); Drug: Placebo

INTERVENTIONS:
Drug: E2/DRSP (BAY 86-4891) dose 1 (SH T04984E) — Single dose administration of E2 + DRSP as a tablet
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: E2/DRSP (BAY 86-4891) dose 2 (80458739) — Single dose administration of E2 + DRSP as a tablet
  Arms: Arm 3; Arm 4; Arm 5; Arm 6
Drug: E2/DRSP (BAY 86-4891) dose 3 (80458755) — Single dose administration of E2 + DRSP as a tablet
  Arms: Arm 3; Arm 4
Drug: E2/DRSP (BAY 86-4891) dose 4 (80458720) — Single dose administration of E2 + DRSP as a tablet
  Arms: Arm 4; Arm 6
Drug: E2/DRSP (BAY 86-4891) dose 5 (80458712) — Single dose administration of E2 + DRSP as a tablet
  Arms: Arm 5; Arm 6
Drug: DRSP (ZK 30595) dose 1 (SH T04984F) — Single dose administration of DRSP as a tablet
  Arms: Arm 1; Arm 2; Arm 4
Drug: DRSP (ZK 30595) dose 2 (80458690) — Single dose administration of DRSP as a tablet
  Arms: Arm 6
Drug: Placebo — Placebo administration in each arm

SUMMARY:
The study will be performed as a multi-center, randomized, double-blind, parallel-group trial in fertile women aged between 18 and 35 years inclusive. A total of 600 volunteers will be randomized into one of the six treatment groups. The study will be performed only in Germany. The investigational drug is an oral contraceptive. It contains the estrogen estradiol (E2) and the progestogen drospirenone (DRSP). As the contraceptive efficacy has not yet been proven for these new regimens, even a protection against unwanted pregnancies cannot be assured. The treatments will be applied daily for 7 cycles of 28 days each without pill-free interval, i.e., for 196 consecutive days. Treatment will be initiated after a screening period of approximately 1 to 2 weeks, the latter focused on confirmation of the baseline safety status. Tablet intake will start on the first day of the first menstrual/withdrawal bleeding after Visit 2, regardless of whether the volunteer is a first user (starter) or switching from another COC. In the following cycles, tablet intake is not to be triggered by any bleeding events. The primary objective of this study is to evaluate and compare the cycle control and bleeding patterns of six different treatment regimens with E2/DRSP during administration for 7 treatment cycles. Volunteers will be provided with a diary to document the intake of study medication, any bleeding events, and days without bleeding, pregnancy test results. Safety will be also assessed. During the whole study period, 4 visits are planned. At Screening and Final examination, a thorough physical examination and a gynecological examination (including breast palpation and cervical smear ) will be performed. Blood samples will be taken for safety laboratory parameters.Additional examinations can be performed any time, if this becomes necessary for medical reasons. At Visit 3 or in case of premature discontinuation of study the investigator will discuss options for follow-up contraception with the volunteer. The volunteer can start the intake of a post-treatment OC on the day after the last tablet intake of study medication, after a negative urine ß-HCG test (home pregnancy test) result.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Age: 18 - 35 years (inclusive), smokers must not be older than 30 years at inclusion
* History of regular cyclic menstrual periods (with a cycle length between 25 and 35 days)
* Willingness to use barrier methods of contraception (condoms with spermicide, diaphragms with spermicide, spermicidal vaginal suppositories) or abstinence during the trial

Exclusion Criteria:

* Pregnancy, lactation (less than three menstrual cycles before Visit 1 following delivery, abortion, or lactation) - Obesity (BMI > 30.0 kg/m2)
* Abnormal, suspicious or unclear cervical smear (a cervical smear has to be taken at Visit 1 or a normal result has to be documented within the last 6 months before Visit 1)
* Laboratory values outside inclusion range at Screening - Any disease that may worsen under hormonal treatment or might interfere with the conduct of the study or the interpretation of the results, as e.g.: - Cardiovascular -- presence or a history of venous or arterial thrombotic/thromboembolic events (e.g., deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident, including prodromi (e.g., transient ischemic attack, angina pectoris) and conditions which could increase the risk to suffer from any of the above mentioned disorders, e.g., a family history indicating a hereditary predisposition. -- uncontrolled arterial hypertension (repeated measurements of systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg)
* Liver -- presence or history of liver tumor (benign or malignant) -- presence or history of severe hepatic disease as long as liver function values have not returned to normal -- jaundice and/or pruritus related to cholestasis -- history of cholestatic jaundice associated with pregnancy or previous COC use
* Metabolic diseases -- uncontrolled diabetes mellitus with vascular involvement severe dyslipoproteinemia
* Other diseases: any known or suspected malignant or premalignant disease, uncontrolled thyroid disorder, chronic inflammatory bowel disease, severe renal insufficiency or acute renal failure, hemolytic uremic syndrome, sickle cell anemia, porphyria, history of hypertriglyceridemia-associated Pancreatitis, systemic lupus erythematodes, pemphigoid gestationis during a previous pregnancy, Sydenham chorea, herpes gestationis, otosclerosis-related hearing loss, history of migraine with focal neurologic symptoms, epilepsy, current or history of clinically significant depression, hereditary angioedema
* Additional sex steroids, other hormonal contraceptive methods (oral, transdermal) during treatment (blister in use at randomization should be finished); intra-uterine devices (IUD) with or without hormone release within 1 month prior to Visit 1, implants within 1 month prior Visit 1, depot progestins within 6 months prior to Visit 1 - Surgical interventions scheduled in the study period

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 635 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of intracyclic bleeding episodes during cycles 2 to 7 | 168 days

SECONDARY OUTCOMES:
Number of intracyclic bleeding days (including spotting) in Cycles 2 to 7 | 168 days
Number of withdrawal bleeding episodes in Cycles 1 to 6 | 168 days
Bleeding pattern | Approximately 7 months
  Bleeding pattern was determined by: - Number of bleeding/spotting days - Number of bleeding days (excluding spotting) - Number of spotting-only days - Number, mean length, maximum length, and range of length of bleeding/spotting episodes - Number, mean length, maximum length, and range of length of spotting-only episodes
Cycle control | Approximately 7 months
  Withdrawal bleeding - Number of volunteers with/without withdrawal bleeding; - Length, maximum intensity, and onset of withdrawal bleeding episodes Intracyclic bleeding (including/excluding spotting) - Number of volunteers with/without intracyclic bleeding; - Number, maximum length, maximum intensity (including spotting only) of intracyclic bleeding episodes - Number of intracyclic bleeding days - Number of volunteers with at least one intracyclic bleeding (including/excluding spotting) episode in Cycles 2 - 6 and in Cycles 2 - 7
Subjective assessment of treatment | Day 196 - Day 210
  The treatment satisfaction assessment was done through a questionaire. The investigator handed it over to the subject and the subject was asked to answer all questions by herself.
Number of participants with adverse events | Approximately 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- Germany (17):
  - Krumbach, Bavaria
  - Nuremberg, Bavaria
  - Hamburg, Hamburg
  - Dietzenbach, Hesse
  - Frankfurt am Main, Hesse
  - Fulda, Hesse
  - Mühlheim am Main, Hesse
  - Dippoldiswalde, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Wurzen, Saxony
  - Blankenburg, Saxony-Anhalt
  - Burg, Saxony-Anhalt
  - Jessen, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Gera, Thuringia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/